CLINICAL TRIAL: NCT01761370
Title: Intragastric Balloon for Treatment of Non Alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D/05/338
Record Dates: First submitted 2011-11-01; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2011-10

CONDITIONS: Non Alcoholic Steatohepatitis
Keywords: Non alcoholic Steatohepatitis; Intra-gastric balloon
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Active Comparator): AHA diet plus exercise with BIB placement
  Interventions: Procedure: AHA diet plus exercise with BIB placement
- Sham control (Sham Comparator): AHA diet plus exercise with sham BIB placement
  Interventions: Procedure: AHA diet plus exercise with sham BIB placement

INTERVENTIONS:
Procedure: AHA diet plus exercise with BIB placement — AHA diet plus exercise with BIB placement for 6 months
  Arms: Treatment
Procedure: AHA diet plus exercise with sham BIB placement — AHA diet plus exercise with sham BIB placement
  Arms: Sham control

SUMMARY:
The study will determine the feasibility of using Bioenteric intragastric balloon (BIB) in the treatment of patients with Non alcoholic Steatohepatitis (NASH).

DETAILED DESCRIPTION:
The Bio-enteric Intra-gastric balloon (BIB) has been shown to be an effective treatment for weight reduction in obese patients. This study will determine the feasibility of using BIB in the treatment of patients with Non alcoholic Steatohepatitis (NASH). It will evaluate the efficacy of the BIB in improving histology of NASH in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 21-65 years of age,
* Had histological evidence of NASH,
* Had a BMI of greater than 27kg/m2, and
* Had failed at least 6 month trial of medical therapy for weight reduction.

Exclusion Criteria:

* Patients with any organic disease of the upper GI tract,
* Were receiving anti-inflammatory drugs,
* Anticoagulants or steroids, or
* Had a history of alcoholism or drug addiction. A hiatus hernia of > 5 cm, an active gastric or duodenal ulcer, and prior or intestinal surgery were considered contraindications to the placement of BIB.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Change in liver histology | 6 months
  The primary outcome measure was liver histology before and after treatment. Assessment of disease activity was done with the use of the NAS, which grades steatosis, lobular inflammation and hepatocellular ballooning.

CONTACTS AND LOCATIONS:
Overall Officials: Yin Mei Lee, MBChB, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore